CLINICAL TRIAL: NCT01450917
Title: Diaphragmatic Height Index: the New Diagnostic Test for Phrenic Nerve Dysfunction
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: Si442/2552(EC2)
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Respiratory Paralysis
MeSH Terms: conditions — Respiratory Paralysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Brachial plexus injured patients with phrenic nerve dysfunction
- Group B: Brachial plexus injured patients without phrenic nerve dysfunction
- Group C: Non brachial plexus injured patients

SUMMARY:
Diaphragmatic contraction is controlled by phrenic nerve which consists of anterior rami of 3rd- 5th cervical nerve roots. Usually, It can't be evaluated from history taking and physical examination. Thus the diaphragmatic elevation on chest radiograph is assumed to identify the phrenic nerve dysfunction. Normally, the right diaphragm is higher than the left side about 1.5 ± 0.9 centimeters or 0.5 ± 0.3 time of vertebral height. Although there are several methods to determine the diaphragmatic elevation from previous studies, the accuracy, reliability, intra and inter-observer variation are problem.

Neurotization is the effective procedure to restore upper extremity function in root avulsion type. Phrenic nerve is one of the common donor nerves which used for this procedure. But sometimes, concomitant injury of this nerve can occur. Therefore, the investigators established "Diaphragmatic height index (DHI)" from chest radiograph to use as the diagnostic test for phrenic nerve dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Brachial plexus injured patients who underwent the neurotization in our institute between 2005-2008
* Non brachial plexus injured patients who underwent the other orthopedic operation in our institute between April-June 2009

Exclusion Criteria:

* Concomitant pneumothorax and/or hemothorax
* Concomitant pulmonary contusion
* Previous pulmonary disease
* Chest wall deformity
* Thoracic or thoracolumbar scoliosis (>10 degrees)
* Hepatomegaly
* Incomplete data

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 220 brachial plexus injured patients who underwent the neurotization and 80 non-brachial plexus injury patients who underwent the orthopaedic operation were retrospectively reviewed. With using nerve electrical stimulator (Aesculap Nerve Stimulator GN 24, Tuttlingen, Germany), in neurotization procedures, phrenic nerve dysfunction is defined by no any diaphragmatic contraction was observed intraoperatively. The enrolled patients were classified into three main groups: (A) BPI patients with phrenic nerve dysfunction group, (B) BPI patients with normal phrenic nerve function group and (C) non-BPI patients group. In group A and B, we further subgroubed into: (1) for the right and (2) for the left side.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2009-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The cut-off point of DHI for diagnosis of phrenic nerve dysfunction | upto 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Saichol Wongtrakul, MD, Principal Investigator — Mahidol University